CLINICAL TRIAL: NCT00396656
Title: A Randomized, Open-label, Multicenter, Cross-over Trial to Evaluate the Efficacy of a 20 Week Treatment of Valsartan 320 mg Versus Atenolol 100 mg in Combination With Hydrochlorothiazide on Microcirculation in Hypertensive Patients
Brief Title: Safety and Efficacy of Valsartan vs Atenolol and Hydrochlorothiazide Combination on Blood Flow in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Anna Mitchell, MD, University Hospital Essen, Essen, Germany et al.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631BDE06
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: hypertension; valsartan; atenolol; hydrochlorothiazide; microcirculation; arterial compliance; pulse wave analysis
MeSH Terms: conditions — Hypertension | interventions — Atenolol; Hydrochlorothiazide; Valsartan

ARMS (2):
- Valsartan followed by atenolol + hydrochlorothiazide (HCTZ) (Experimental): After a 2-week washout period, patients were treated with valsartan for 20 weeks followed by one week in which it was tapered off. Patients received valsartan 160 mg for 4 weeks, followed by valsartan 320 mg for 16 weeks. The valsartan dose was then tapered off to 80 mg for one week. Patients took valsartan film coated tablets orally once a day (od) in the morning.
  After a second 2-week washout period, patients were treated with atenolol plus HCTZ for 20 weeks. Patients received atenolol 100 mg for 20 weeks. Patients took atenolol tablets orally once a day (od) in the morning. Patients received HCTZ 12.5 mg for 4 weeks starting at the beginning of the 5th week and then received 25 mg for 12 weeks. Patients took HCTZ tablets orally once a day (od) in the morning.
  Interventions: Drug: Atenolol; Drug: Hydrochlorothiazide (HCTZ)); Drug: Valsartan
- Atenolol + hydrochlorothiazide (HCTZ) followed by valsartan (Experimental): After a 2-week washout period, patients were treated with atenolol plus HCTZ for 20 weeks followed by one week in which atenolol was tapered off and HCTZ was discontinued. Patients received atenolol 100 mg for 20 weeks. Patients took atenolol tablets orally once a day (od) in the morning. Patients received HCTZ 12.5 mg for 4 weeks starting at the beginning of the 5th week and then received 25 mg for 12 weeks. Patients took HCTZ tablets orally once a day (od) in the morning.
  After a second 2-week washout period, patients were treated with valsartan for 20 weeks. Patients received valsartan 160 mg for 4 weeks, followed by valsartan 320 mg for 16 weeks. Patients took valsartan film coated tablets orally once a day (od) in the morning.
  Interventions: Drug: Atenolol; Drug: Hydrochlorothiazide (HCTZ)); Drug: Valsartan

INTERVENTIONS:
Drug: Atenolol — 100 mg tablets orally once a day (od) in the morning.
Drug: Hydrochlorothiazide (HCTZ)) — 12.5 or 25 mg tablets orally once a day (od) in the morning.
Drug: Valsartan — 80 mg, 160 mg, or 320 mg tablets orally once a day in the morning

SUMMARY:
This study evaluated the effect of valsartan on small vessel blood flow in patients with mild-to-moderate hypertension in direct comparison to atenolol and hydrochlorothiazide.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian; male or female outpatients and age between 40-65 years of age, inclusive.
* At Visit 2 all patients must have a mean sitting diastolic blood pressure (msSBP) of ≥ 90 mmHg and < 110 mmHg.

Exclusion Criteria:

* If a single reading for arterial hypertension in msSBP > 180 mmHg or msDBP > 110 mmHg at any visit after randomization.
* Inability to discontinue all prior antihypertensive medications safely for a period of 2 weeks prior to randomization.
* Known history of hypotensive symptoms or orthostatic hypotension.
* Concomitant use of statins or statin intake during the four weeks prior to Visit 1.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* A history of heart failure (NYHA II-IV).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma Ag, Principal Investigator — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharma Ag, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: First Treatment Period
Arm/Group | Valsartan Followed by Atenolol + Hydrochlorothiazide (HCTZ) | Atenolol + Hydrochlorothiazide (HCTZ) Followed by Valsartan
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Treatment Period
Arm/Group | Valsartan Followed by Atenolol + Hydrochlorothiazide (HCTZ) | Atenolol + Hydrochlorothiazide (HCTZ) Followed by Valsartan
Started | 15 | 13
Completed | 15 | 12
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes patients that received valsartan followed by atenolol + hydrochlorothiazide and patients that received atenolol + hydrochlorothiazide followed by valsartan.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Post-treatment Microcirculation at Acetylcholine (ACH) Injected Sites Compared to NaCl Injected Sites
Description: 10 µl of acetylcholine (ACH) at 3 concentrations (10-7, 10-8, 10-9 M) was injected intra-dermally at 3 sites on the forearms. NaCl was injected at 2 sites on the forearms. Microcirculation was measured using laser doppler velocimetry before and 12 times in the 30 minutes following injection. The mean difference of the 12 post-injection measurements to the pre-injection measurement was calculated. Means for the 3 ACH and the 2 NaCl sites were calculated and compared. Microcirculation was measured in perfusion units which is an arbitrary measure specific to each laser doppler scanner.
Time Frame: At end of each treatment period (Week 21 and Week 43)
Population: Intent-to-treat (ITT) population: All randomized patients with at least one valid post-baseline primary efficacy measurement in both treatment periods.
Measure: Mean (Standard Deviation); unit: Perfusion units
Groups:
- Valsartan: Patients received valsartan 160 mg for 4 weeks, followed by valsartan 320 mg for 16 weeks. The valsartan dose was then tapered off to 80 mg for one week. Patients took valsartan film coated tablets orally once a day (od) in the morning.
- Atenolol + Hydrochlorothiazide: Patients received atenolol 100 mg for 19 weeks. In the last week of this intervention, the atenolol dose was reduced to 50 mg. Patients took atenolol tablets orally once a day (od) in the morning. Patients received hydrochlorothiazide 100 mg for 15 weeks starting at the beginning of the 5th week of this intervention. In the last week of this intervention, the hydrochlorothiazide dose was increased to 25 mg. Patients took hydrochlorothiazide tablets orally once a day (od) in the morning.
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Number analyzed (Participants) | 27 | 27
Perfusion units | 61.21 (38.11) | 61.04 (49.16)

2. Secondary Outcome: Difference in Mean Post-treatment Microcirculation at Acetylcholine (ACH) Plus L-NMMA Injected Sites Compared to NaCl Injected Sites
Description: 10 µl of acetylcholine (ACH) at 3 concentrations (10-7, 10-8, 10-9 M) plus 10 µl L-NMMA (10-6 M) was injected intra-dermally at 3 sites on the forearms. NaCl was injected at 2 sites. Microcirculation was measured using laser doppler velocimetry before and 12 times in the 30 minutes following injection. The mean difference of the 12 post-injection measurements to the pre-injection measurement was calculated. Means for the 3 ACH and the 2 NaCl sites were calculated and compared. Microcirculation was measured in perfusion units which is an arbitrary measure specific to each laser doppler scanner.
Time Frame: At end of each treatment period (Week 21 and Week 43)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Number analyzed (Participants) | 27 | 27
Perfusion units | -9.11 (22.19) | -5.60 (40.47)

3. Secondary Outcome: Difference in Mean Post-treatment Microcirculation at a Sodium Nitroprusside Injected Site Compared to NaCl Injected Sites
Description: 10 µl of sodium nitroprusside at a concentration of 10-7 M was injected intra-dermally at 1 site on the forearms. NaCl was injected at 2 sites on the forearms. Microcirculation was measured using laser doppler velocimetry before and 12 times in the 30 minutes following injection. The mean difference of the 12 post-injection measurements to the pre-injection measurement was calculated. A mean for the 2 NaCl sites was calculated and compared to the sodium nitroprusside mean. Microcirculation was measured in perfusion units which is an arbitrary measure specific to each laser doppler scanner.
Time Frame: At end of each treatment period (Week 21 and Week 43)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Number analyzed (Participants) | 27 | 27
Perfusion units | 120.65 (74.52) | 128.14 (63.79)

4. Secondary Outcome: Mean Post-treatment Microcirculation at NaCl Injected Sites
Description: 10 µl of NaCl was injected intra-dermally at 2 sites on the forearms. Microcirculation was measured using laser doppler velocimetry before and 12 times in the 30 minutes following injection. The mean difference of the 12 post-injection measurements to the pre-injection measurement was calculated. A mean for the 2 NaCl sites was calculated. Microcirculation was measured in perfusion units which is an arbitrary measure specific to each laser doppler scanner.
Time Frame: At end of each treatment period (Week 21 and Week 43)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Number analyzed (Participants) | 27 | 27
Perfusion units | 44.78 (47.53) | 50.96 (67.88)

5. Secondary Outcome: Arterial Pressure Waveform Augmentation Index at the End of Treatment
Description: Using applanation tonometry, the arterial pulse form measured at the wrist was analyzed using computerized pulse wave analysis. The arterial pressure waveform has two components; the first is the forward traveling wave when the left ventricle contracts and the second is the reflected wave returning from the periphery. The augmentation index is the ratio of the first and second systolic peaks and is used as a surrogate measure of arterial stiffness.
Time Frame: At end of each treatment period (Week 21 and Week 43)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Number analyzed (Participants) | 27 | 27
Ratio | 139.05 (20.64) | 144.51 (21.97)

6. Secondary Outcome: Arterial Pressure Waveform Pulse Wave Velocity at the End of Treatment
Description: Using applanation tonometry, the arterial pulse form measured at the wrist was analyzed using computerized pulse wave analysis. The arterial pressure waveform has two components; the first is the forward traveling wave when the left ventricle contracts and the second is the reflected wave returning from the periphery. Pulse wave velocity is the speed of the forward traveling wave and can be used as a measure of arterial stiffness since the more rigid the wall of the artery, the faster the wave moves.
Time Frame: At end of each treatment period (Week 21 and Week 43)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Number analyzed (Participants) | 27 | 27
Meters per second | 8.07 (1.28) | 7.60 (1.18)

ADVERSE EVENTS:
Description: Two patients in the treatment sequence atenolol + hydrochlorothiazide followed by valsartan did not receive treatment during the second treatment period and were excluded from the valsartan safety population analysis set.
Arm/Group | Valsartan | Atenolol + Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/30
Other Adverse Events (participants affected / at risk) | 16/28 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan (N=28) | Atenolol + Hydrochlorothiazide (N=30)
Diverticulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan (N=28) | Atenolol + Hydrochlorothiazide (N=30)
Vertigo (Ear and labyrinth disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 6
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.